CLINICAL TRIAL: NCT03229772
Title: Demonstration of the "SPECT/CT System With CZT Detectors" Imaging Performance in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 117.02-2015-GES-0002
Record Dates: First submitted 2016-05-11; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects indicated for dynamic nuclear medicine scanning (Other): The trial will consist of a single arm composed of subjects with preexisting indications for dynamic nuclear medicine scanning at the site. All patients will undergo nuclear medicine scintigraphy using the GE Discovery 670 NM/CT device with and without CZT enabled during a single visit.
  Interventions: Device: Discovery NM/CT 670 CZT Imaging Scan

INTERVENTIONS:
Device: Discovery NM/CT 670 CZT Imaging Scan — At a single visit, subjects will undergo nuclear medicine scintigraphy imaging scanning on the investigational GE Discovery 670 NM/CT CZT (with CZT) device and the commercial GE Discovery 670c (without CZT).

SUMMARY:
The primary purpose of the study is to obtain sample clinical images that are evaluated by physicians in support of regulatory submissions. Additionally, the study will provide data for current and future product development and it will provide clinical images and data for marketing use.

ELIGIBILITY:
Inclusion Criteria:

1. are 18-years old and older;
2. is able to sign and date the informed consent form; AND
3. have been prescribed by a physician a nuclear medicine exam that is within the intended use of the device.

Exclusion Criteria:

1. Patients who were referred for dynamic nuclear medicine scan because of the need to be injected twice (once for the conventional acquisition and once for the investigational device) that would result in an increase dose burden on patient.
2. Pregnant or lactating women
3. Who were previously enrolled in this study;
4. Who have contraindication for the radiopharmaceutical
5. Who have any conditions that, in the opinion of the Investigator, would interfere with the evaluation of the results or constitute a health hazard for the subject;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic Image Quality | 12 weeks
  Diagnostic Image Quality will be rated by 2 radiologist using a 5 point Likert Scale
Image Resolution | 12 weeks
  Image Resolution will be rated by 2 radiologist using a 5 point Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Keidar, MD, Principal Investigator — Rambam Health Care Center
Locations (1):
- Rambam Health Care Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No